CLINICAL TRIAL: NCT00652314
Title: Evaluation of an Absorbable Surgical Hemostatic Agent: Thrombi-Gel® Versus Gelfoam-Thrombin
Acronym: Control
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vascular Solutions LLC (Industry)
Collaborators: King Pharmaceuticals is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0307; The CONTROL Study (Other: Vascular Solutions)
Record Dates: First submitted 2008-03-28; First posted 2008-04-03 (Estimated); Results first posted 2016-03-07 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2016-02

CONDITIONS: Operation Site Bleed
Keywords: Hemostatic products; Surgical hemostasis; Thrombi-gel; Gelatin Sponge; Time to hemostasis
MeSH Terms: interventions — Gelatin Sponge, Absorbable

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 - Thrombi-gel treatment (Experimental): Thrombi-gel treatment
  Interventions: Device: Thrombi-Gel
- 2 - Gelatin Sponge (Gelfoam) (Active Comparator): Gelatin Sponge (Gelfoam) plus thrombin
  Interventions: Device: Thrombi-Gel

INTERVENTIONS:
Device: Thrombi-Gel — Applicaton of Hemostatic product during surgery
  Other Names: Gelatin Sponge (Gelfoam) plus thrombin

SUMMARY:
This trial is designed as a prospective, multi-center, randomized, feasibility clinical trial to evaluate the safety and efficacy of Thrombi-Gel as an absorbable surgical hemostat.

Within this clinical evaluation, Thrombi-Gel will be compared to the current standard of care, a gelatin sponge (Gelfoam) plus Thrombin JMI, by using a 2:1 randomization ratio. Subjects will be randomized to one of two (2) treatment groups. One (1) group will be treated with Thrombi-Gel, while one (1) group will be treated with the gelatin sponge plus thrombin. All study data will be analyzed according to the subjects' assigned randomization group assignment, regardless of the treatment actually delivered.

DETAILED DESCRIPTION:
This is a prospective, randomized, multi-center investigation with a minimum of seventy five (75) study subjects designed to evaluate the safety and effectiveness of the Thrombi-Gel product as an absorbable hemostat in the surgical patient population.

Subjects who are undergoing orthopedic/spinal, general, cardiac, hepatic or vascular surgical procedures should be considered for this investigation. Subjects can be pre-screened utilizing standard of care data for the specified inclusion/exclusion criteria to ensure that they are eligible for treatment in the investigation. If the subject appears to qualify for the investigation, the subject will then be asked to give his/her written informed consent. If, during surgery, the surgeon encounters a bleeding site that he or she is unable or unwilling to easily control due to failure or impracticality of conventional methods (sutures and/or cautery), the subject may be enrolled and randomized to receive either the investigational or control treatment. If the subject has multiple bleeding sites, each site to a maximum of 5 sites, may be treated with the assigned surgical hemostat. However, only the first site treated will be used to determine study objectives. All subjects will be followed through their hospitalization.

A follow-up evaluation will be conducted at approximately 30 and 60 days post-procedure to determine the long-term effectiveness of the hemostatic treatment received, incidence of late adverse events, and interim immunologic response to the study treatment device. Follow-up evaluations will include obtaining a blood specimen that evaluates for antibody development, coagulation, and Factor Va testing. Blood samples will be sent to independent labs for analysis.

From baseline to the final study exam, data pertaining to the investigational objectives will be recorded on the appropriate case report forms at the predetermined study intervals. The investigation will be conducted at a minimum of five (5) sites, but no more than fifteen (15) sites.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is 18 years of age or older
2. The subject is undergoing an orthopedic/spinal, general, cardiac, hepatic, or vascular surgical procedure (neurosurgical, ophthalmic or urological procedures must be excluded)
3. The subject is willing and able to provide appropriate informed consent
4. The subject is willing and able to comply with the requirements of the study protocol, including the predefined follow-up evaluations

Inclusion criteria to be determined during the surgical procedure:

1. The subject has an intraoperative bleeding site which the surgeon is unable or unwilling to easily control with conventional methods (cautery, sutures)

Exclusion Criteria:

1. The subject is known or suspected to be pregnant (verified in a manner consistent with institution's standard of care), or is lactating
2. The subject has a known allergy to bovine derived products or any other materials used in the Thrombi-Gel product
3. The subject has an active infection at the surgical site
4. The use of hemostatic agents are contraindicated for the subject
5. The subject has a known bleeding disorder (including thrombocytopenia [< 100,000 platelet count], thrombobasthenia, hemophilia, or von Willebrand disease)
6. The subject has received antibiotic solutions/powders at the intended application site
7. The subject has had surgery at the intended application site ≤ 6 months before the current surgical procedure
8. The subject is unavailable for follow-up
9. The subject is currently participating in another investigational device or drug trial
10. The subject has previously participated in this trial (Protocol 0307) or the Thrombi-Paste trial (Protocol 0507)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2008-03; Primary Completion 2009-10 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Dolan, MD, Principal Investigator — Lahey Clinic
Locations (7):
- United States (7):
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Lahey Clinic, Burlington, Massachusetts
  - Michigan Vascular Research Center, Flint, Michigan
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Sanford Clinic, Sioux Falls, South Dakota
  - Southwest Regional Clinical Research, Lubbock, Texas
  - Texas Tech University Health Sciences Center, Lubbock, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- 2 - Gelatin Sponge (Gelfoam) Plus Thrombin: Gelatin Sponge (Gelfoam) plus thrombin
  Thrombi-Gel: Applicaton of Hemostatic product during surgery
Period: Overall Study
Arm/Group | 1 - Thrombi-gel Treatment | 2 - Gelatin Sponge (Gelfoam) Plus Thrombin
Started | 62 | 35
Completed | 53 | 26
Not Completed | 9 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 - Thrombi-gel Treatment | 2 - Gelatin Sponge (Gelfoam) Plus Thrombin | Total
Number analyzed (Participants) | 62 | 35 | 97
Age, Customized [Number; unit: participants]
  >= to 18 Years | 62 | 35 | 97
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 21 | 58
  Male | 25 | 14 | 39

OUTCOME MEASURES:

1. Primary Outcome: The Primary Objective of This Investigation is to Gather Information to Support the Effectiveness of Thrombi-Gel as Compared to a Gelatin Sponge (Gelfoam) Plus Thrombin as an Adjunct to Hemostasis in Multi-specialty Surgical Settings.
Description: Evaluation for hemostasis began immediately following application of the safety product. Hemostasis assessments were to be made every minute for the first 10 minutes post application. If hemostasis was not observed within 10 minutes, the treatment site was to be monitored and the research teams were asked to record the specific number of minutes until hemostasis was observed.
Time Frame: Time to hemostasis (minutes)
Measure: Mean (Standard Deviation); unit: Time to hemostasis (minutes)
Arm/Group | 1 - Thrombi-gel Treatment | 2 - Gelatin Sponge (Gelfoam) Plus Thrombin
Number analyzed (Participants) | 62 | 35
Time to hemostasis (minutes) | 4.01 (4.15) | 3.72 (4.75)

2. Secondary Outcome: Effectiveness: Device Success (Defined as the Number of Subjects With First Bleeding Site Applications for Which Hemostasis Was Obtained Within 6 Minutes of Study Device Application Without the Need for Adjunctive Treatment)
Time Frame: Procedure, up to 6 minutes post procedure
Measure: Number; unit: participants
Arm/Group | 1 - Thrombi-gel Treatment | 2 - Gelatin Sponge (Gelfoam) Plus Thrombin
Number analyzed (Participants) | 62 | 35
participants | 50 | 29

3. Secondary Outcome: Effectiveness: Hemostatic Handling Characteristics (Surgeon's Questionnaire)
Description: Ease of application to bleeding site as assessed by surgeon questionnaire for hemostatic handling characteristics.
Time Frame: Procedure (application through end of procedure)
Population: Note that the number of participants analyzed (62 and 33) applies to each set of five rows below which apply to the following categories: Ease of application to bleeding site, conformance to tissue surfaces, ease of delivery to hard to reach surfaces, and ease of preparation for use.
Measure: Number; unit: participants
Arm/Group | 1 - Thrombi-gel Treatment | 2 - Gelatin Sponge (Gelfoam) Plus Thrombin
Number analyzed (Participants) | 62 | 33
participants
  Ease of application to bleeding site - 1 (easy) | 57 | 29
  Ease of application to bleeding site - 2 | 5 | 4
  Ease of application to bleeding site - 3 | 0 | 0
  Ease of application to bleeding site - 4 | 0 | 0
  Ease of application to bleeding site - 5 (hard) | 0 | 0
  Conformance to tissue surfaces - 1 (well) | 47 | 28
  Conformance to tissue surfaces - 2 | 15 | 4
  Conformance to tissue surfaces - 3 | 0 | 1
  Conformance to tissue surfaces - 4 | 0 | 0
  Conformance to tissue surfaces - 5 | 0 | 0
  Ease of delivery to hard to reach surfaces-1(easy) | 38 | 24
  Ease of delivery to hard to reach surfaces - 2 | 14 | 5
  Ease of delivery to hard to reach surfaces - 3 | 3 | 1
  Ease of delivery to hard to reach surfaces - 4 | 0 | 0
  Ease of delivery to hard to reach surfaces-5(hard) | 0 | 0
  Ease of preparation for use - 1 (easy) | 56 | 24
  Ease of preparation for use - 2 | 4 | 3
  Ease of preparation for use - 3 | 2 | 6
  Ease of preparation for use - 4 | 0 | 0
  Ease of preparation for use - 5 | 0 | 0

4. Secondary Outcome: Safety: Incidence Rate of Device-related Adverse Events
Time Frame: Procedure, up to 60 days post procedure
Measure: Number; unit: participants
Arm/Group | 1 - Thrombi-gel Treatment | 2 - Gelatin Sponge (Gelfoam) Plus Thrombin
Number analyzed (Participants) | 62 | 35
participants
  Serious | 2 | 0
  Non-Serious | 1 | 0

5. Secondary Outcome: Safety: Immunological Testing for Factor Va Antibodies and Coagulation Parameters
Time Frame: 0 day, 30 day, and 60 days post procedure
Measure: Number; unit: participants
Arm/Group | 1 - Thrombi-gel Treatment | 2 - Gelatin Sponge (Gelfoam) Plus Thrombin
Number analyzed (Participants) | 62 | 35
participants
  Bovine FV/Va (0 Day) | 11 | 3
  Bovine FV/Va (30 Day) | 17 | 9
  Bovine FV/Va (60 Day) | 11 | 7
  Bovine Thrombin (0 Day) | 12 | 4
  Bovine Thrombin (30 Day) | 15 | 7
  Bovine Thrombin (60 Day) | 14 | 4
  Human FV/Va (0 Day) | 9 | 7
  Human FV/Va (30 Day) | 12 | 10
  Human FV/Va (60 Day) | 10 | 5
  Human Thrombin (0 Day) | 3 | 2
  Human Thrombin (30 Day) | 7 | 3
  Human Thrombin (60 Day) | 4 | 3

ADVERSE EVENTS:
Time Frame: 60-Day
Description: Adverse events reviewed by an independent clinical events committee (CEC).
Arm/Group | 1 - Thrombi-gel Treatment | 2 - Gelatin Sponge (Gelfoam) Plus Thrombin
Serious Adverse Events (participants affected / at risk) | 11/62 | 5/35
Other Adverse Events (participants affected / at risk) | 33/62 | 22/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 - Thrombi-gel Treatment (N=62) | 2 - Gelatin Sponge (Gelfoam) Plus Thrombin (N=35)
Abnormal Thrombosis (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Hematoma (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Infection/Abscess (Infections and infestations) | 2 (3) | 1 (1)
Other (General disorders) | 6 (7) | 4 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 - Thrombi-gel Treatment (N=62) | 2 - Gelatin Sponge (Gelfoam) Plus Thrombin (N=35)
Foreign Body / Hypersensitivity Reaction / Allergic Reaction (Immune system disorders) | 1 (1) | 2 (2)
Infection/Abscess (Infections and infestations) | 1 (1) | 1 (1)
Other (General disorders) | 32 (68) | 22 (56)
Tissue Necrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less